CLINICAL TRIAL: NCT00448370
Title: Role of Placenta Growth Factor in Sickle Acute Chest Syndrome
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CCHMC 06-09-57; R01 (Other Grant/Funding Number: HL079916)
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Anemia, Sickle Cell
Keywords: Anemia, sickle cell
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to find out whether Placenta Growth Factor (PlGF) and related tests can predict the development of acute chest syndrome (ACS) in patients with sickle cell disease (SCD) during a period where patients are well and during admission to the hospital for an acute sickle event to see if these measures can predict the development of ACS. Understanding events precipitating ACS may lead to preventative and interventional therapies which will improve patient outcomes and quality of life.

DETAILED DESCRIPTION:
The proposed research is a clinical study designed to test the hypothesis that PlGF levels in blood at baseline in patients with SCD will correlate with leukotriene (LT) levels and will be reflective of the degree of airway obstruction; and that acute elevations in PlGF levels will occur during an acute sickle event and precede clinical and radiological recognition of ACS. This is a biological study that does not fall into the criteria of a phase I-IV trial.

Measurements will be done at two stages. First, patients who are admitted to the hospital with an acute sickle event will have a daily evaluation for the first 4 days of the admission or up until the patient has an ACS event. Measurements of inpatient spirometry (at primary site only) and impulse oscillometry will be performed daily. Measurements on 35 ACS events with ACS developing on the 3rd/4th day of admission will be collected. Measurements on patients developing ACS will be compared to those who do not develop ACS will allow for earlier prediction of ACS. Finally, patients who have an ACS or admission for an acute sickling event will be evaluated again after 3-4 weeks in order to get a baseline measurement. One hundred baseline measurements will be made. Twenty of these baseline patients will also have one or two additional baseline evaluations at subsequent clinic visits to evaluate the overall non-event baseline distribution and intra-subject baseline variability. Patients will have measurements repeated if admitted for an acute event greater than one year since the last baseline measurement . These measurements will be used to see if there is any prognostic information for a subsequent acute or ACS event. Some patients may only have baseline data collected.

ELIGIBILITY:
Inclusion criteria:

1. Patients must have a diagnosis of SCD (HbSS, HbSC or HbS beta/thal) by hemoglobin electrophoresis or gene mapping. Very few patients with HbSC or HbS beta/thal would go onto develop ACS, but they will serve as important controls.
2. Patients must be ≥5.5 years of age and ≤30 years of age.
3. Patients must be able to comply with pulmonary function tests.

Exclusion criteria:

1. Patients taking anti-leukotriene medications such as montelukast (Singulair®) or zileuton (Zyflo®) 30 days prior to enrollment will be ineligible, although patients with SCD and asthma who are not on leukotriene inhibitors will be eligible.
2. Patients with known congenital heart disease or with congenital lung abnormality/disease that will affect the pulmonary function testing and methacholine challenge testing will be ineligible (examples include patients with cyanotic heart disease, immotile cilia syndrome, cystic fibrosis, diaphragmatic hernia).
3. Any patient with neurologic abnormalities, stroke, developmental delay, or other medical condition that would preclude cooperation with pulmonary function testing or compliance with protocol procedures will be ineligible.
4. Patients over 30 years of age will be ineligible.
5. Patients who are pregnant or nursing.
6. Patients on chronic transfusions will be ineligible.

   * If patients come off transfusion therapy, they will be eligible 3 months following the last transfusion.
   * Patients receiving simple transfusions will be eligible, but baseline measurements will be made 3 months following the simple transfusion.

Ages: 66 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will have sickle cell disease (HbSS, HbSC, or Hb Sbeta-thalassemia) and will be equal to or greater than 5.5 years old.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2007-03; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes in plasma PlGF levels and urine LT levels in SCD patients | Baseline and serially through the development of an Acute Sickle Event

SECONDARY OUTCOMES:
Relationship of clinical parameters of severity of SCD and circulating levels of PlGF, leukotrienes, proinflammatory cytochemokines and pulmonary function tests | Baseline and serially through the development of an Acute Sickle Event

CONTACTS AND LOCATIONS:
Overall Officials: Karen Kalinyak, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Punam Malik, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- See also: Cincinnati Children's Hospital Medical Center — http://cincinnatichildrens.org
- See also: Cincinnati Comprehensive Sickle Cell Center — http://www.cincinnatichildrens.org/svc/alpha/b/blood/programs/sickle-cell